CLINICAL TRIAL: NCT01712763
Title: Treatment With Long Acting GnRH Antagonist Degarelix in Women With Endometriosis Recurrence
Brief Title: Degarelix in the Treatment of Endometriosis Recurrence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre for Endocrinology and Reproductive Medicine, Italy (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C06/2012
Record Dates: First submitted 2012-10-18; First posted 2012-10-24 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2022-02

CONDITIONS: Endometriosis
Keywords: Endometriosis; long acting GnRH antagonist; Degarelix; Recurrence; Pelvic Pain
MeSH Terms: conditions — Endometriosis; Recurrence; Pelvic Pain | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Leuprolide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Degarelix (Experimental): 180 women will be treated with degarelix 120mg in one administration
  Interventions: Drug: degarelix
- leuprolide acetate 11.25 mg/ml (Active Comparator): 180 women will be treated with leuprolide acetate 11.25 mg/ml only once covering three months
  Interventions: Drug: Leuprolide Acetate 11.25 MG/ML (Enantone 11,25)

INTERVENTIONS:
Drug: degarelix — 180 women will be treated with degarlix 120 mg, in only one administration covering three months
  Other Names: firmagon
  Arms: Degarelix
Drug: Leuprolide Acetate 11.25 MG/ML (Enantone 11,25) — 180 women will be treated with leuprolide acetate11.25 only once covering three months
  Other Names: Enantone 11.25
  Arms: leuprolide acetate 11.25 mg/ml

SUMMARY:
The long acting GnRH antagonist degarelix will be tested for the treatment of women with endometriosis recurrence compared with classical GnRH analog treatment. Pain symptom disappearance and disease free time during follow-up will be the outcomes for establishing which medical treatment is the best in endometriosis recurrence treatment.

DETAILED DESCRIPTION:
Endometriosis is a chronic disease affecting 5-10% of women in reproductive age, showing recurrence after surgery at least in 20-50% after 5 years of follow-up. The long acting GnRH antagonist degarelix, which do not have the flare-up effect at the opposite of GnRH agonist and strongly suppress LH secretion and thecal cell activity may show a better effects on endometrial implants than GnRH agonist.

ELIGIBILITY:
Inclusion Criteria:

* women affected by endometriosis showing recurrence of pain symptoms
* previous surgery for endometriosis

Exclusion Criteria:

* presence of other systemic diseases

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2012-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
disease free time | 24 months
  time without pain symptoms due to the disease recurrence

SECONDARY OUTCOMES:
time of disappearance pain | 24 months
  time needed during treatment to improve the pain symptoms

OTHER OUTCOMES:
reduction of endometriosis lesions | 24 months
  endometriosis lesions regression during treatment evidenced by MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: MARCO SBRACIA, MD, Study Chair — Centre for Endocrinology and Reproductive Medicine, Italy
Locations (3):
- Albania Spitali Amerikan, Tirana, Albania
- Nadezda Women's Health Hospital, Sofia, Bulgaria
- Cerm-Hungaria, Rome, Italy